CLINICAL TRIAL: NCT06711172
Title: Assessing the Feasibility of a Whole Health Coaching Intervention for Veterans With Chronic Multisymptom Illness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: War Related Illness and Injury Study Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1592308
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chronic Multisymptom Illness
Keywords: Health coaching, chronic multisymptom illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Coaching (Experimental)
  Interventions: Other: Health coaching intervention

INTERVENTIONS:
Other: Health coaching intervention — The health coaching intervention will consist of seventeen, 30 to 60-minute telehealth sessions that were dispersed over six months. Participants will work closely with a health coach to create a plan for making appropriate lifestyle changes and for accomplishing the clinical recommendations that were received from their comprehensive evaluation at the War Related Illness and Injury Study Center.

SUMMARY:
This study examines the impact of a clinical whole health coaching program aimed at improving Veteran's health and well-being by promoting engagement/adherence with clinical recommendations and increasing healthy lifestyle behaviors in treatment-seeking Veterans receiving care at the DC and CA War Related Illness and Injury Study Centers.

ELIGIBILITY:
Inclusion Criteria:

•Veterans receiving a clinical evaluation at the War Related Illness and Injury Study Centers in Washington, DC or Palo Alto, California.

Exclusion Criteria:

* Current active suicidal or homicidal ideation
* Current or lifetime history of a psychiatric disorder with primary psychotic features
* Current or lifetime bipolar disorder
* Acute or unstable psychiatric condition(s) and/or chronic illnesses that would benefit from immediate referral for treatment
* Neurological disorders such as Alzheimer's disease, advanced Parkinson's disease, and unstable epilepsy
* Pregnancy
* Current exposure to trauma, or exposure to trauma in the past 3 months
* Current or within the past 30 days substance abuse or dependence (except nicotine)
* Excessive alcohol intake defined as an AUDIT score ≥ 4 for men and an AUDIT score ≥ 3 for women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment rate) | Through study completion, an average of 6 months
  Calculated as the number of participants who consented into the study divided by the number of participants who were approached for study participation.
Feasibility (retention rate) | Through study completion, an average of 6 months
  Calculated as a percentage for each time point (3 months and 6 months).
Feasibility (adherence rate) | Through study completion, an average of 6 months
  Calculated as the number of health coaching sessions completed out of 17 total sessions.
Safety of a health coaching intervention | Through study completion, an average of 6 months
  Reported as the number of adverse events self-reported by participants during the intervention
Acceptability | Through study completion, an average of 6 months
  Acceptability was evaluated qualitatively using feedback captured during health coaching sessions.

SECONDARY OUTCOMES:
RAND 36-Item Health Survey (SF-36) | Baseline to 3 months and baseline to 6 months
  To measure physical and mental health-related quality of life.
Personal Health Inventory (PHI) | Baseline to 3m and baseline to 6m
  The PHI is a 15-item, self-assessment questionnaire that assesses the eight self-care areas identified in the VA's Whole Health, "Circle of Health."
Pittsburgh Sleep Quality Index (PSQI) | Baseline to 6 months
  To assess sleep quality and sleep disturbances
Generalized Anxiety Disorder scale (GAD-7) | Baseline to 6 months
  To assess the level of anxiety symptoms
VA Pain Numeric Pain Rating Score | Baseline to 6 months
  To assess pain levels
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline to 6 months
  To evaluate mindfulness
Patient Health Questionnaire-8 (PHQ8) | Baseline to 6 month
  To assess the level of depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca McCullers, RN, NBC-HWC, Principal Investigator — War Related Illness and Injury Study Center
Locations (1):
- Washington, DC Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No